CLINICAL TRIAL: NCT04400994
Title: The Use of IVIG in Combination With Rituximab VS Rituximab as the First Line Treatment of Pemphigus
Brief Title: IVIG With Rituximab vs Rituximab as First Line Treatment of Pemphigus
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Sze-Man Wong, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW19-671
Record Dates: First submitted 2020-04-27; First posted 2020-05-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pemphigus
Keywords: Pemphigus; intravenous immunoglobulins; rituximab
MeSH Terms: conditions — Pemphigus | interventions — Rituximab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rituximab only (Active Comparator): * Rituximab infusion 375mg/m2 body surface area (BSA) weekly for 4 weeks from baseline (week 0, 1, 2, 3)
  * Rituximab infusion 375mg/m2 BSA weekly for 4 weeks at week 24 (week 24, 25, 26, 27)
  * Rituximab infusion 375mg/m2 BSA weekly for 2 weeks at week 52 (week 52, 53)
  * Rituximab infusion 375mg/m2 BSA weekly for 4 weeks at week 76 (week 76, 77)
  * A total of 12 doses of rituximab will be given in 55 weeks
  Interventions: Drug: Rituximab
- Rituximab and IVIG (Experimental): * Rituximab (375 mg/m2 BSA) once a week for 4 weeks (week 1, 2, 3);
  * Week 4: Rituximab + IVIG 2g per kg
  * Week 5, 6, 7: Above treatment repeated for 2nd cycle, infusion of rituximab (375 mg/m2 BSA) once a week for 4 weeks (week 5, 6, 7);
  * Week 8: Rituximab + IVIG 2g/kg
  * In months 3, 4, 5, 6, patients received a single infusion of rituximab (375 mg/m2 BSA) plus infusion of 2g/kg IVIG
  * Thus in 6-month period patients received a total of 12 infusions of rituximab and 7 infusions of IVIG
  * If a patient was clinically free of disease at end of 6 months, additional infusions of IVIG will be given at week 30, 38, 48, 60 and 76
  * A total of 12 doses of rituximab and 12 cycles of IVIG will be given
  Interventions: Drug: Rituximab; Other: IVIg

INTERVENTIONS:
Drug: Rituximab — Rituximab would be given intravenously.
  * IV Rituximab is prediluted at a dose of 500mg in 500ml of 0.9% normal saline (i.e. 1:1 dilution, 1 mg/ml)
  * Initial infusion rate starts at a rate of 50mg/hr (50ml/hr)
  * If no hypersensitivity/anaphylaxis reaction occurs, increase infusion rate in 50mg/hr (50 ml/hr) increments every 30 minutes
  * Maximum infusion rate is 400 mg/hr (400 ml/hr)
  * Subsequent infusion: start at rate of 100mg/hr (100 ml/hr), increase 100mg/hr (100 ml/hr) increments every 30 minutes
  * Monitor temperature, BP HR, respiratory rate and SpO2 every 30 minutes
  Other Names: MabThera
Other: IVIg — IVIg would be given in combination with Rituximab intravenously. Infusion plan of IVIg:
  0 min: 50ml/hour 15 min: 75ml/hour 30 min: 100ml/hour 45 min: 125ml/hour 60 min: 150ml/hour 75 min & beyond: 180ml/hour
  Other Names: Privigen
  Arms: Rituximab and IVIG

SUMMARY:
Pemphigus is a rare acquired autoimmune disease in which immunoglobulin G (IgG) antibodies target desmosomal proteins to produce intraepithelial, and mucocutaneous blisters. It is potentially fatal and the average mortality of pemphigus vulgaris (PV) was 75% before the introduction of corticosteroids in the early 1950s.

Traditionally, treatment of pemphigus included high dose systemic corticosteroids with or without adjuvant immunosuppressants. However; the prolonged use of high dose steroids carries significant side effects. A recent randomized trial has proved the efficacy of Rituximab, a monoclonal anti-CD20 antibody against B-lymphocytes, as an efficacious therapy for pemphigus. Early use of rituximab was associated with better clinical outcomes, hence combination treatment of rituximab and intravenous immunoglobulins (IVIG) has shown to be effective for refractory pemphigus cases and can potentially induce long-term complete remission and lower risks infectious complications.

In this study, investigators will evaluate the efficacy and safety of early use of rituximab with or without IVIG in patients with moderate to severe pemphigus using protocols that were similar to those previously published, investigators will also aim to measure the impact of health care economics and in doing so, assess the cost and benefits of both treatment arms.

DETAILED DESCRIPTION:
Pemphigus is a rare acquired autoimmune disease in which immunoglobulin G (IgG) antibodies target desmosomal proteins to produce intraepithelial, and mucocutaneous blisters. It is potentially fatal and the average mortality of pemphigus vulgaris (PV) was 75% before the introduction of corticosteroids in the early 1950s.

Traditionally, treatment of pemphigus included high dose systemic corticosteroids with or without adjuvant immunosuppressants. However; the prolonged use of high dose steroids carries significant side effects. A recent randomized trial has proved the efficacy of Rituximab, a monoclonal anti-CD20 antibody against B-lymphocytes, as an efficacious therapy for pemphigus. Furthermore, early use of rituximab was associated with associated with better clinical outcomes. Moreover, combination treatment of rituximab and intravenous immunoglobulins (IVIG) has shown to be effective for refractory pemphigus cases and can potentially induce long-term complete remission and lower risks infectious complications.

Cost effectiveness is an important issue and while combination of IVIG and rituximab has been advocated, the cost of such treatment is substantial and whether it poses any benefit over rituximab alone, or with other more conventional immunosuppressive agents, has not been established. Both treatment approaches have been previously published in high impact journals.

In this study, investigators aim to evaluate the efficacy and safety of early use of rituximab with or without IVIG in patients with moderate to severe pemphigus using protocols that were similar to those previously published. Apart from complete remission and adverse effects, investigators will also aim to measure the impact of health care economics and in doing so, assess the cost and benefits of both treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from patient
* Ages Eligible for Study: 18 years to 75 years (Adult, Older Adult)
* Newly or recently diagnosed (less than 18 months) diagnosed pemphigus vulgaris or pemphigus foliaceus based on clinical features; histological features of acantholysis via skin or mucosal biopsy; and intercellular staining pattern of indirect immunofluorescence or serological detection of DSG 1 or DSG 3 by enzyme-linked immunosorbent assay (ELISA)
* Moderate to severe active disease, as defined by overall PDAI >= 15 or skin involvement BSA>= 5%. 9 [Annex 1]
* Receiving standard-of-care oral prednisolone up to 1.5 mg/kg/day
* Women who are sexually active and not postmenopausal, agreement to remain abstinent or use 2 effective methods of contraception.
* Ability to comply with study protocol as deemed by investigator's assessment

Exclusion criteria:

* Age <18 or >75
* Pregnant women or nursing mother
* Already diagnosed pemphigus patients diagnosed > 18 months
* Non-consenting patients, or patient who cannot be followed up regularly
* Patient with history of serious allergy or anaphylactic reaction to monoclonal antibody treatment
* Severe heart failure (NYHA Class III or IV)
* Unstable angina or myocardiac infarction within last 3 months or post-infarction heart failure
* Anaemia (haemoglobin <10g/dL), Neutropenia (<1000/mm3), Lymphopenia (<900/mm3), thrombocytopenia (<100,000/mm3)
* Renal insufficiency eGFR <60
* Liver insufficiency of ALT/ALT > 2 times normal limit range
* Positive test results for hepatitis C (HCV) serology at screening *Patients who are HepBs Ag positive, or HepBs Ag negative and anti-HepBc Ab - positive: Patients who are HepBs Ag positive - will be started on entecavir 0.5mg daily, and will be referred to a gastroenterologist for further follow up.

Patients who are HepBs Ag negative, and HBc Ab positive, with detectable HepB DNA levels - will be started on entecavir 0.5mg daily, and will be referred to a gastroenterologist for further follow up.

Patients who are HepBs Ag negative, HBc Ab positive, with no detectable HepB DNA levels - will be started on entecavir 0.5mg daily, and will be continued on entecavir for at least 18 months after completion of last dose of rituximab.

* Blood test positive for HIV
* Signs of active infection on CXR
* Positive interferon gamma release assay Quantiferon or T.Spot TB test: must be treated with at least 4 weeks post initiation of isoniazid or other TB therapy
* Inherited or acquired severe immunodeficiency
* History of malignancy
* Patient with active severe infection (excluding fungal infections of the nail), which has required antibiotic treatment within 2 week prior to study enrolment
* Infection requiring hospitalisation or intravenous antibiotic treatment within the last 8 weeks prior to enrolment
* Past history of osteomyelitis, or fasciitis, septic arthritis within the last one year
* Patients with drug induced pemphigus. A thorough medication history will be taken to rule out drug induced pemphigus including D-penicillamine, angiotensin-converting enzyme inhibitors, angiotensin receptor blockers and cephalosporins
* Evidence of any new or uncontrolled concomitant disease that in the investigators' judgement would preclude the patients participation
* Patients with history of allergy or adverse events to IVIG or rituximab treatment10
* Treatment with intravenous immunoglobulins, plasmaphoresis within the last 8 weeks prior to randomization
* Previous treatment with rituximab or any monoclonal antibody inducing profound lymphopenia
* Treatment with live or attenuated vaccine within the last 28 days prior to randomization

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
relapse-free complete remission | From baseline up to 208 weeks
  Percentage of participants who achieve relapse-free complete remission

SECONDARY OUTCOMES:
Time to protocol defined disease flare | From baseline up to 208 weeks
  Time to protocol defined disease flare
Duration of complete remission | From baseline up to 208 weeks
  Duration of complete remission, evaluated by the PDAI activity score
Number of protocol defined disease flares | From baseline up to 208 weeks
  Number of protocol defined disease flares
Time to initial complete remission | From baseline up to 208 weeks
  Time to initial complete remission, evaluated by the PDAI activity score
Change in health-related quality of life: Dermatology Life Quality Index (DLQI) Score | Baseline, Week 4, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192
  Change in health-related quality of life as measured by the Dermatology Life Quality Index (DLQI) Score.
  The DLQI is calculated by summing the score of each question resulting in maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Occurrence of severe treatment adverse events | Baseline, week 4, 12, 24, 36, 48, 60, 72, 96, 120, 144, 168, 192
  Safety endpoints: Occurrence of treatment adverse events, serious adverse events (grade 3 or 4) based on common terminology criteria for adverse events (CTCAE). Death from any cause. Adverse events leading to discontinuation, vital signs, and laboratory tests
Blood DSG 1 and 3 levels | Baseline week 0, week 4, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192
  Blood DSG 1 and 3 levels
Blood lymphocyte level (CBC) | Baseline week 0, week 4, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192
  Blood lymphocyte level (CBC)
Blood CD19/20 mean B cell counts percentage | Week 0, week 4, 12, 24, 36, 48, 60, 72, 84, 96, 120, 144, 168, 192
  Blood CD19/20 mean B cell counts percentage
Number of rescue therapy given | Baseline up to Week 208
  Number of rescue therapy given

CONTACTS AND LOCATIONS:
Overall Officials: Sze Man Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, Central, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harman KE, Brown D, Exton LS, Groves RW, Hampton PJ, Mohd Mustapa MF, Setterfield JF, Yesudian PD. British Association of Dermatologists' guidelines for the management of pemphigus vulgaris 2017. Br J Dermatol. 2017 Nov;177(5):1170-1201. doi: 10.1111/bjd.15930. No abstract available. PMID 29192996
- [Background] Hertl M, Jedlickova H, Karpati S, Marinovic B, Uzun S, Yayli S, Mimouni D, Borradori L, Feliciani C, Ioannides D, Joly P, Kowalewski C, Zambruno G, Zillikens D, Jonkman MF. Pemphigus. S2 Guideline for diagnosis and treatment--guided by the European Dermatology Forum (EDF) in cooperation with the European Academy of Dermatology and Venereology (EADV). J Eur Acad Dermatol Venereol. 2015 Mar;29(3):405-14. doi: 10.1111/jdv.12772. Epub 2014 Oct 22. PMID 25338479
- [Background] Joly P, Maho-Vaillant M, Prost-Squarcioni C, Hebert V, Houivet E, Calbo S, Caillot F, Golinski ML, Labeille B, Picard-Dahan C, Paul C, Richard MA, Bouaziz JD, Duvert-Lehembre S, Bernard P, Caux F, Alexandre M, Ingen-Housz-Oro S, Vabres P, Delaporte E, Quereux G, Dupuy A, Debarbieux S, Avenel-Audran M, D'Incan M, Bedane C, Beneton N, Jullien D, Dupin N, Misery L, Machet L, Beylot-Barry M, Dereure O, Sassolas B, Vermeulin T, Benichou J, Musette P; French study group on autoimmune bullous skin diseases. First-line rituximab combined with short-term prednisone versus prednisone alone for the treatment of pemphigus (Ritux 3): a prospective, multicentre, parallel-group, open-label randomised trial. Lancet. 2017 May 20;389(10083):2031-2040. doi: 10.1016/S0140-6736(17)30070-3. Epub 2017 Mar 22. PMID 28342637
- [Background] Lunardon L, Tsai KJ, Propert KJ, Fett N, Stanley JR, Werth VP, Tsai DE, Payne AS. Adjuvant rituximab therapy of pemphigus: a single-center experience with 31 patients. Arch Dermatol. 2012 Sep;148(9):1031-6. doi: 10.1001/archdermatol.2012.1522. PMID 22710375
- [Background] Ahmed AR, Spigelman Z, Cavacini LA, Posner MR. Treatment of pemphigus vulgaris with rituximab and intravenous immune globulin. N Engl J Med. 2006 Oct 26;355(17):1772-9. doi: 10.1056/NEJMoa062930. PMID 17065638
- [Background] Feldman RJ, Christen WG, Ahmed AR. Comparison of immunological parameters in patients with pemphigus vulgaris following rituximab and IVIG therapy. Br J Dermatol. 2012 Mar;166(3):511-7. doi: 10.1111/j.1365-2133.2011.10658.x. Epub 2012 Jan 19. PMID 21967407
- [Background] Ahmed AR, Kaveri S. Reversing Autoimmunity Combination of Rituximab and Intravenous Immunoglobulin. Front Immunol. 2018 Jul 18;9:1189. doi: 10.3389/fimmu.2018.01189. eCollection 2018. PMID 30072982
- [Background] Ahmed AR, Nguyen T, Kaveri S, Spigelman ZS. First line treatment of pemphigus vulgaris with a novel protocol in patients with contraindications to systemic corticosteroids and immunosuppressive agents: Preliminary retrospective study with a seven year follow-up. Int Immunopharmacol. 2016 May;34:25-31. doi: 10.1016/j.intimp.2016.02.013. Epub 2016 Feb 23. PMID 26919279
- [Background] Boulard C, Duvert Lehembre S, Picard-Dahan C, Kern JS, Zambruno G, Feliciani C, Marinovic B, Vabres P, Borradori L, Prost-Squarcioni C, Labeille B, Richard MA, Ingen-Housz-Oro S, Houivet E, Werth VP, Murrell DF, Hertl M, Benichou J, Joly P; International Pemphigus Study Group. Calculation of cut-off values based on the Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) and Pemphigus Disease Area Index (PDAI) pemphigus scoring systems for defining moderate, significant and extensive types of pemphigus. Br J Dermatol. 2016 Jul;175(1):142-9. doi: 10.1111/bjd.14405. Epub 2016 Apr 3. PMID 26800395
- [Background] US Department of Health and Human Services, National Institutes of Health, National Cancer Institute. Common terminology criteria for Adverse Events (CTCAE), version 5.0: Nov 27, 2017.
- [Background] Murrell DF, Pena S, Joly P, Marinovic B, Hashimoto T, Diaz LA, Sinha AA, Payne AS, Daneshpazhooh M, Eming R, Jonkman MF, Mimouni D, Borradori L, Kim SC, Yamagami J, Lehman JS, Saleh MA, Culton DA, Czernik A, Zone JJ, Fivenson D, Ujiie H, Wozniak K, Akman-Karakas A, Bernard P, Korman NJ, Caux F, Drenovska K, Prost-Squarcioni C, Vassileva S, Feldman RJ, Cardones AR, Bauer J, Ioannides D, Jedlickova H, Palisson F, Patsatsi A, Uzun S, Yayli S, Zillikens D, Amagai M, Hertl M, Schmidt E, Aoki V, Grando SA, Shimizu H, Baum S, Cianchini G, Feliciani C, Iranzo P, Mascaro JM Jr, Kowalewski C, Hall R, Groves R, Harman KE, Marinkovich MP, Maverakis E, Werth VP. Diagnosis and management of pemphigus: Recommendations of an international panel of experts. J Am Acad Dermatol. 2020 Mar;82(3):575-585.e1. doi: 10.1016/j.jaad.2018.02.021. Epub 2018 Feb 10. PMID 29438767
- [Background] Liu KSH, Seto WK, Lau EHY, Wong DK, Lam YF, Cheung KS, Mak LY, Ko KL, To WP, Law MWK, Wu JT, Lai CL, Yuen MF. A Territorywide Prevalence Study on Blood-Borne and Enteric Viral Hepatitis in Hong Kong. J Infect Dis. 2019 May 24;219(12):1924-1933. doi: 10.1093/infdis/jiz038. PMID 30668746
- [Background] Seto WK, Chan TS, Hwang YY, Wong DK, Fung J, Liu KS, Gill H, Lam YF, Lie AK, Lai CL, Kwong YL, Yuen MF. Hepatitis B reactivation in patients with previous hepatitis B virus exposure undergoing rituximab-containing chemotherapy for lymphoma: a prospective study. J Clin Oncol. 2014 Nov 20;32(33):3736-43. doi: 10.1200/JCO.2014.56.7081. Epub 2014 Oct 6. PMID 25287829
- [Background] Tsai YF, Yang CI, Du JS, Lin MH, Tang SH, Wang HC, Cho SF, Liu YC, Su YC, Dai CY, Hsiao HH. Rituximab increases the risk of hepatitis B virus reactivation in non-Hodgkin lymphoma patients who are hepatitis B surface antigen-positive or have resolved hepatitis B virus infection in a real-world setting: a retrospective study. PeerJ. 2019 Sep 9;7:e7481. doi: 10.7717/peerj.7481. eCollection 2019. PMID 31565551